CLINICAL TRIAL: NCT05602441
Title: Living Together With Chronic Disease: Informal Support for Diabetes Management in Vietnam
Brief Title: Living Together With Chronic Disease: Informal Support for Diabetes Management in Vietnam (VALID)
Acronym: VALID
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Thai Binh University of Medicine and Pharmacy (Other)
Collaborators: University of Copenhagen (Other); University of Southern Denmark (Other)
Responsible Party: Principal Investigator, Thanh Duc Nguyen, Associate professor, Head of Health mangement Department, Thai Binh University of Medicine and Pharmacy
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: VALID
Record Dates: First submitted 2022-09-15; First posted 2022-11-02 (Actual); Last update posted 2022-11-02 (Actual); Status verified 2022-10

CONDITIONS: Diabete Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Intervention Model Description: Pilot intervention study with pre- and post assessment of effects
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- VALID - diabetes supportive clubs (Experimental): VALID - diabetes supportive clubs
  Interventions: Behavioral: VALID - diabetes supportive clubs

INTERVENTIONS:
Behavioral: VALID - diabetes supportive clubs — The VALID - diabetes supportive clubs comprised diabetes classes and diabetes clubs, to highlight two prominent aspects of diabetes self-management: education and peer support.
  The diabetes club meeting was held twice a month during a 9-month intervention, consisting of a focused delivery of the knowledge and discussion following the topic in the monthly class. Club meetings also included dedicated time for blood glucose testing and sharing experiences to deal with the difficulties of the periodic insurance examinations process. Finally, the club meetings provided the participants with emotional support to deal with the stigma and sadness in their daily lives.
  Core messages aimed to strengthen daily self-management and boost the spiritual bond between individuals with T2D toward a healthy, happy life with T2DM. In addition, the intervention aimed to strengthen the capacities of grassroots health care workers in diabetes consultations and communication in rural communities.

SUMMARY:
Insufficient self-management is a significant barrier for people with type 2 diabetes (T2D) to achieve glycemic control and reduce the risk of acute and long-term diabetes complications which negatively affect the quality of life and increase the risk of diabetes-related death. This pre-post study aimed to evaluate the impact of a peer-based club intervention to improve self-management among people living with T2D in two rural communities in Vietnam.

DETAILED DESCRIPTION:
Vietnam has up to 3.9 million people diagnosed with T2D. This situation poses challenges for Vietnam's long-term health services, where the healthcare workforce is currently deficient compared to the practical needs and having an imbalanced geographical distribution of the health workforce, especially highly specialized practitioner staff, between urban and rural areas. The majority of primary care settings - community health centers are incapable of diagnosis, treatment, or follow-up management of diabetes patients due to lack of qualified human resources, medications, and advanced medical equipment. Informal support from non-professionals plays an essential role among people with T2D and potentially assists with optimal diabetes self-management. An additional widely acknowledged type of non-professional supporter is the community health worker. Therefore, to boost the advantages and address the disadvantages of peer and VHW support for enhanced diabetes self-management capability in the rural communities, an intervention conducted in Vietnam's Thai Binh province as part of the larger interdisciplinary project, Living Together with Chronic Disease: Informal Support for Diabetes Management in Vietnam (VALID) (grant number 17-M09-KU), was developed.

Study aim The present pre-and post-study aimed to test the feasibility of a peer support intervention after one year of implementation, emphasizing the impact of diabetes clubs on T2DM self-management in two rural communities in Thai Binh, Vietnam.

Methods Study design An intervention with a pre-post study was implemented between January 2021 and January 2022. Pre- and post-intervention data were collected following a structured questionnaire and a clinical examination.

Setting The study was conducted in Thai Binh province with a population of 1.86 million people.

Due to two COVID-19 lockdown periods, the intervention, including diabetes classes and clubs, had to be put on hold for one month in May and November 2021.

The investigators organized a participatory design workshop in 2019 to discuss in detail with people with T2D participating in the qualitative study, a part of the project, and VHW, thus, developing a culturally appropriate intervention for diabetes self-management. Based on the findings that manifested in the obstacles and a strong desire for knowledge and peer support in self-management among people with T2D in rural communities, the investigators designed a diabetes management intervention, "Living healthy and well with diabetes," including diabetes classes and diabetes clubs, to highlight two prominent aspects of diabetes self-management: education and peer support. Moreover, due to the limited availability of comprehensive and attractive health education communication materials on diabetes, the investigators decided to develop a new set of diabetes educational materials. The investigators also introduced the concept of representative patients (RPs), those who lived with long-term T2D while also being active in their communities and open about their disease. 30 VHWs and 32 RPs from eighteen villages in two rural communities participated in "train-the-trainer" classes held once a month for nine months developed by the investigators. The training topics focused on diabetes self-management principles and blood glucose fluctuations prevention and treatment on special occasions.

Before and after each diabetes class, VHWs and RPs organized and moderated interactive diabetes learning clubs with other patients in their villages who were willing to participate. The diabetes club meeting was held twice a month during a 9-month intervention, consisting of a focused delivery of the knowledge and discussion following the topic in the monthly class. Club meetings also included dedicated time for blood glucose testing and sharing experiences to deal with the difficulties of the periodic insurance examinations process. Finally, the club meetings provided the participants with emotional support to deal with the stigma and sadness in their daily lives.

Core messages aimed to strengthen daily self-management and boost the spiritual bond between individuals with T2D toward a healthy, happy life with T2DM.

Sampling To compare the pre-post proportion of statistical power of 90%, a two-sided level of significance of 5%, equal group sizes, the anticipated proportion in the baseline population of 65%, and to detect a difference in proportions of -0.15 between the two groups (test - reference group), should include at least 237 people.

Ethics of research Ethical clearance was approved by the Medical Ethics Committee of Thai Binh University of Medicine and Pharmacy, Vietnam (decision 11/2018, 23rd November 2018). Every participant was informed about the purpose of the study, that participation was voluntary, and signed the written consent before participating in the examination and interview. Participants could withdraw at any time from the study. The participants were checked-up at the commune healthcare centers and interviewed in their homes. The completed questionnaires were managed and stored securely at Thai Binh University of Medicine and Pharmacy, Vietnam.

ELIGIBILITY:
Inclusion Criteria:

* Individuals diagnosed with or treated for T2D over 18 years old
* Residing in two selected communes
* Without acute and/or severe illness
* Able to answer the questionnaire completely
* Agreed to participate voluntarily
* Participated in both pre - post-study and the intervention program.

Exclusion Criteria:

* Refusal to continue participating in study
* Migration
* Illness or hospitalization

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 229 (Actual)
Dates: Start 2021-01-12 (Actual); Primary Completion 2022-01-11 (Actual); Study Completion 2023-05-31 (Estimated)

PRIMARY OUTCOMES:
Change in glycated haemoglobin from baseline to 12 months post intervention | Baseline and 12 months post intervention
  HbA1c goal for adults is 7 % or less

SECONDARY OUTCOMES:
Change in medication adherence -Morisky Medication Adherence Scale-8 (MMAS-8) from baseline | Start intervention and 12 months post intervention
  The total score ranged from 0 to 8 and was classified into three degrees of Medication adherence, including low (<6 points), medium (6 - <8 points), and high (8 points)
Change in body mass index - BMI from baseline | Baseline and 12 months post intervention
  Body mass index (BMI) was calculated using the Asia-Pacific classification based on the formula of (weight (kg)/ [height (m)2
Change in mental health Self Reporting Questionnaire 20-Item (SRQ-20) from baseline | Baseline and 12 months post intervention
  The clinical reference index of SRQ-20 is 7, where a score exceeding 7 is considered to reflect emotional pain.
Change in systolic blood pressure from baseline | Baseline and 12 months post intervention
  The systolic blood pressure (BP) reading were obtained with the left arm at the heart level using an automatic digital blood pressure monitor (Omron, Japan)
Change in diastolic blood pressure from baseline | Baseline and 12 months post intervention
  The diastolic blood pressure (BP) reading were obtained with the left arm at the heart level using an automatic digital blood pressure monitor (Omron, Japan)
Change in quality of life measured by Short Form-36 (SF36) from baseline | Baseline and 12 months post intervention
  The SF-36 consists of eight scaled scores, which are the weighted sums of the questions in their section. To score the SF-36, scales are standardized with a scoring algorithm or by the SF-36v2 scoring software to obtain a score ranging from 0 to 100. Higher scores indicate better health status.A mean score of 50 has been articulated as a normative value.
change in awareness of hypo-/hyperglycemia from baseline | Baseline and 12 months post intervention
  Ad hoc developed questions
Change in self-management of diabetes from baseline | Baseline and 12 months post intervention
  Measured by ad hoc developed questions ad hoc developed questions
Change in knowledge and practices of foot care from baseline | Baseline and 12 months post intervention
  Measured by hoc developed questions
Change in tobacco smoking habit from baseline | Baseline and 12 months post intervention
  Measured by hoc developed questions
Change in alcohol consumption from baseline | Baseline and 12 months post intervention
  Measured by hoc developed questions
Change in unmet need of support of relevance for type 2 diabetes management from baseline | Baseline and 12 months post intervention
  Measured by hoc developed questions
Change in diabetes distress measured by Diabetes Distress - Screening Scale 17 (DDS-17) from baseline | Baseline and 12 months post intervention
  The scale yields an overall distress score based on the average responses on the 1-6 scale for all 17 items. A mean question score of 3 or higher (moderate distress) indicate a level of distress worthy. Low score indicate low distress level.Lowest means score is 1 and highest possible mean score is 6.

CONTACTS AND LOCATIONS:
Locations (1):
- Thai Binh University of Medicine and Pharmacy, Thái Bình, Vietnam

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Dang NT, Phong Vu T, M Gammeltoft T, Christian Bygbjerg I, W Meyrowitsch D, Sondergaard J. Pre-/-post-analyses of a feasibility study of a peer-based club intervention among people living with type 2 diabetes in Vietnam's rural communities. PLoS One. 2023 Nov 28;18(11):e0290355. doi: 10.1371/journal.pone.0290355. eCollection 2023. PMID 38015901